CLINICAL TRIAL: NCT02516592
Title: A 12-week Treatment, Multi-center, Randomized, Double-blind, Double-dummy, Parallel Group Study to Assess the Efficacy and Safety of Switching From Salmeterol/Fluticasone to QVA149 (Indacaterol Maleate/Glycopyrronium Bromide) in Symptomatic COPD Patients
Brief Title: Assessment of Switching From Salmeterol/Fluticasone to Indacaterol/Glycopyrronium in a symtomaticCOPD Patient Cohort
Acronym: FLASH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A3405
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 110/50 micrograms (Experimental): QVA149 110/50 micrograms o.d. Capsules for inhalation
  Interventions: Drug: QVA149 110/50 micrograms
- salmeterol/fluticasone 50/500 micrograms (Active Comparator): salmeterol/fluticasone 50/500 micrograms b.i.d. Dry inhalation powder
  Interventions: Drug: Salmeterol/fluticasone 50/500 microgrammes

INTERVENTIONS:
Drug: QVA149 110/50 micrograms — QVA149 110/50 micrograms o.d. capsules for inhalation, supplied in blisters via a single dose dry powder inhalater (SDDPI)
  Arms: QVA149 110/50 micrograms
Drug: Salmeterol/fluticasone 50/500 microgrammes — Salmeterol/fluticasone 50/500 microgrammes b.i.d.dry inhalation powder delivered via Accuhaler / Diskus device
  Arms: salmeterol/fluticasone 50/500 micrograms

SUMMARY:
This study will investigate whether switching symptomatic COPD patients from a fixed-dose combination of salmeterol/fluticasone 50/500 µg b.i.d. to a fixed dose combination of QVA149 110/50 µg o.d. leads to improved lung function and airflow. It will also assess the effect on symptom burden, breathlessness, and use of rescue medication after this switch.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female ≥ 40 years
* Current or ex-smokers who have a smoking history of at least 10 pack years (Ten pack years are defined as 20 cigarettes per day for 10 years or 10 cigarettes per day for 20 years). An ex-smoker is defined as a patient who has not smoked for ≥ 6 months at visit 1
* Confirmed diagnosis of COPD and post-bronchodilator FEV1 ≥ 30% and < 80% of the predicted normal value and post-bronchodilator FEV1/FVC < 0.70 at visit 1
* Treated with salmeterol/fluticasone 50/500 µg b.i.d. for at least 3 months prior to visit 1
* Documented CAT score of ≥ 10 at Visit 1 and 2

Exclusion Criteria:

* Treatment with any LAMA in the 2 weeks prior to visit 1
* Presence of any contraindication, warning, precaution, hypersensitivity in the approved prescribing information for salmeterol/fluticasone
* Prior or current diagnosis of asthma
* More than one COPD exacerbation requiring treatment with antibiotics and/or systemic corticosteroids and/or hospitalization in the year prior to Visit 1
* Patients who developed a COPD exacerbation of any severity within the 6 weeks before the screening (Visit 1) or between screening (Visit 1) and start of treatment (Visit 2) will not be eligible but will be permitted to be re-screened after a minimum of 6 weeks after the resolution of the COPD exacerbation
* Respiratory tract infection within 4 weeks prior to Visit 1
* Respiratory tract infection between Visit 1 and 2. Patients can be re-screened 4 weeks after resolution of the infection
* Requiring oxygen therapy prescribed for >12 hours per day
* Onset of respiratory symptoms, including a COPD diagnosis prior to age 40 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- Australia (8):
  - Novartis Investigative Site, Coffs Harbour, New South Wales
  - Novartis Investigative Site, Drummoyne, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Cairns, Queensland
  - Novartis Investigative Site, Daw Park, South Austrailia
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Glen Osmond, South Australia
  - Novartis Investigative Site, Murdoch, Western Australia
- Egypt (3):
  - Novartis Investigative Site, Al Fayyum
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- India (5):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Mohali, Punjab
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, New Delhi
- Israel (8):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Tel Giborim, Holon
- Lebanon (5):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Hazmiyeh
  - Novartis Investigative Site, Saida
- Malaysia (6):
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Taiping, Perak
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Miri, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Philippines (5):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, San Pablo City, Laguna
- Saudi Arabia (2):
  - Novartis Investigative Site, Riyadh, SAU
  - Novartis Investigative Site, Jeddah
- South Africa (5):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Gatesville
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Phoenix
- Taiwan (4):
  - Novartis Investigative Site, Kaoshiung
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Erzurum
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Konya
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Trabzon
  - Novartis Investigative Site, Yenisehir/Izmir

REFERENCES:
- [Derived] Frith PA, Ashmawi S, Krishnamurthy S, Gurgun A, Hristoskova S, Pilipovic V, Hamann AM, Backer A, Olsson P, Kostikas K, Diaz DV; FLASH Investigators. Efficacy and safety of the direct switch to indacaterol/glycopyrronium from salmeterol/fluticasone in non-frequently exacerbating COPD patients: The FLASH randomized controlled trial. Respirology. 2018 Dec;23(12):1152-1159. doi: 10.1111/resp.13374. Epub 2018 Aug 3. PMID 30074294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 502 patients were randomized, of which 498 patients were included in the Full Analysis Set (FAS)
Period: Overall Study
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms
Started | 251 | 251
Full Analysis Set | 248 | 250
Completed | 235 | 238
Not Completed | 16 | 13
Not completed — Patient withdrew consent | 5 | 2
Not completed — Protocol deviation | 4 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Patient/guardian decision | 2 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Abnormal test procedure result | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of randomized study medication; patients were analyzed according to the treatment they were randomized to. A total of 502 patients were randomized, of which 498 patients were included in the Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms | Total
Number analyzed (Participants) | 251 | 251 | 502
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The full analysis set (FAS) included all randomized patients who received at least one dose of randomized study medication; patients were analyzed according to the treatment they were randomized to.
  Years
    number analyzed (Participants) | 248 | 250 | 498
    (all) | 65 (9.14) | 65.1 (8.44) | 65 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The full analysis set (FAS) included all randomized patients who received at least one dose of randomized study medication; patients were analyzed according to the treatment they were randomized to.
  Participants
    number analyzed (Participants) | 248 | 250 | 498
    Female | 28 | 26 | 54
    Male | 220 | 224 | 444
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The full analysis set (FAS) included all randomized patients who received at least one dose of randomized study medication; patients were analyzed according to the treatment they were randomized to
  Participants
    number analyzed (Participants) | 248 | 250 | 498
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 115 | 118 | 233
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 0 | 2
    White | 123 | 126 | 249
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Pre-dose FEV1 in Both Arms
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Mean trough pre-dose FEV1 at Week 12 is defined as the average of the measurements taken -45min and -15min pre study medication dose in the clinic after 12 weeks of treatment (Day 84). The baseline measurement is defined as the average of the scheduled FEV1 values prior to first intake of randomized study drug at Day 1 (Visit 2).
Time Frame: Baseline, week 12
Population: The full analysis set (FAS) included all randomized patients who received at least one dose of randomized study medication; patients were analyzed according to the treatment they were randomized to
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms
Number analyzed (Participants) | 248 | 250
Liters | 0.036 (0.0151) | -0.009 (0.0152)
Statistical Analysis 1: Comparison: QVA149 110/50 Micrograms vs Salmeterol/Fluticasone 50/500 Micrograms; Test type: Superiority; p = 0.028, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [0.005 to 0.084]

2. Secondary Outcome: Transitional Dyspnea Index (TDI) Focal Score
Description: Transition Dyspnea Index (TDI) is an instrument used to assess a participant's level of dyspnea. The TDI focal score have three domains: functional impairment, magnitude of task and magnitude of effort. TDI domains were rated from -3 (major deterioration) to 3 (major improvement) and rates summed for transition focal score ranged from -9 to 9; negative scores indicate deterioration. A TDI focal score of ≥1 was defined as a clinically important improvement from baseline.
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms
Number analyzed (Participants) | 248 | 250
Score on a scale | 3.24 (0.405) | 2.79 (0.399)
Statistical Analysis 1: Comparison: QVA149 110/50 Micrograms vs Salmeterol/Fluticasone 50/500 Micrograms; Test type: Superiority; p = 0.063, Mixed Models Analysis; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.03 to 0.94]

3. Secondary Outcome: Change From Baseline in FVC (Forced Vital Capacity)
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. FVC wil follow the same analysis as for FEV1
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms
Number analyzed (Participants) | 248 | 250
Liters | 0.073 (0.0248) | -0.028 (0.0250)
Statistical Analysis 1: Comparison: QVA149 110/50 Micrograms vs Salmeterol/Fluticasone 50/500 Micrograms; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.037 to 0.167]

4. Secondary Outcome: Change From Baseline in Total Symptom Score- CAT (COPD Assessment Test)
Description: The participants will record their COPD symptoms in this test before every clinic visit, this will include : cough, phlegm, chest tightness, breathlessness, limitation in activities, energy, soundly sleep, etc. A higher score indicates a worse health status. The result is immediately available without the need for any calculation, apart from summing the scores on individual items. Scores of 0 - 10 represent mild, 11 - 20 represent moderate, 21 - 30 represent severe and 31 - 40 represent very severe clinical impact of COPD upon the patient.
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms
Number analyzed (Participants) | 248 | 250
Score on a scale | 13.4 (0.48) | 13.8 (0.47)
Statistical Analysis 1: Comparison: QVA149 110/50 Micrograms vs Salmeterol/Fluticasone 50/500 Micrograms; Test type: Superiority; p = 0.319, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.3 to 0.4]

5. Secondary Outcome: Change From Baseline in Mean Daily Use of Rescue Medication
Description: Use of rescue medication (number of puffs taken in the previous 12 hours) is recorded morning and evening, by the patient, in a paper diary. A negative change from baseline indicates an improvement.
Time Frame: over 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | QVA149 110/50 Micrograms | Salmeterol/Fluticasone 50/500 Micrograms
Number analyzed (Participants) | 248 | 250
Number of puffs | 1.05 (0.132) | 1.09 (0.130)
Statistical Analysis 1: Comparison: QVA149 110/50 Micrograms vs Salmeterol/Fluticasone 50/500 Micrograms; Test type: Superiority; p = 0.662, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.20 to 0.13]

ADVERSE EVENTS:
Time Frame: All AEs starting on or after the time of first administration of double-blind study drug but not later than 7 days (30 days in the case of an SAE) after the last administration are included in the summaries
Groups:
- QVA149: QVA149 110/50 micrograms o.d. Capsules for inhalation
- Salm/Flut: salmeterol/fluticasone 50/500 micrograms b.i.d. Dry inhalation powder
Arm/Group | QVA149 | Salm/Flut
All-Cause Mortality (participants affected / at risk) | 1/248 | 1/250
Serious Adverse Events (participants affected / at risk) | 9/248 | 9/250
Other Adverse Events (participants affected / at risk) | 39/248 | 50/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=248) | Salm/Flut (N=250)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Entropion (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Penetrating aortic ulcer (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=248) | Salm/Flut (N=250)
Dry mouth (Gastrointestinal disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Viral upper respiratory tract infection (Infections and infestations) | 3 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypertension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT02516592/SAP_000.pdf
  • Study Protocol (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02516592/Prot_001.pdf